CLINICAL TRIAL: NCT02897258
Title: Thrombosis and Haemorrhage in Chronic Hemodialysis Patients - T2HD
Brief Title: Thrombosis and Haemorrhage in Chronic Hemodialysis Patients
Acronym: T2HD
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, GUILLEMIN Francis, MD, Professor, Central Hospital, Nancy, France
Other Study IDs: T2HD-01
Record Dates: First submitted 2016-08-30; First posted 2016-09-13 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Renal Failure
Keywords: Dialysis; Thrombosis; Haemorrhage
MeSH Terms: conditions — Kidney Failure, Chronic; Thrombosis; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Without anticoagulant/antiplatelet
- Treated with antiplatelet only
- Treated with anticoagulant only
- With antiplatelet/anticoagulant

SUMMARY:
The study T2HD "Thrombosis and Haemorrhage in chronic hemodialysis patients" is a study of pharmacoepidemiology observational, retrospective cohort, multicenter including 12 dialysis centers for adults Lorraine.

The main objective is to :

Describe the prescribing practices of drugs anticoagulants and antiplatelet agents in chronic hemodialysis patients in the Lorraine region.

The second objective is to :

Study the impact of these practices on the survival and the occurrence of major clinical events, thrombotic and hemorrhagic.

DETAILED DESCRIPTION:
All adult patients aged 18 and over who started a new hemodialysis replacement therapy in Lorraine between 01/01/2009 and 31/12/2010 are identified from the registry REIN (Epidemiology and Information Network in nephrology). The latter are included in the study T2HD to the initiation of dialysis and followed until the date point 30/06/2013.

The outcome was survival without major clinical event. Are considered major clinical events: acute coronary syndrome, acute limb ischemia, deep venous thrombosis, arterial thrombosis, pulmonary embolism, thrombosis First, ischemic or hemorrhagic stroke, the digestive hemorrhage, and severe bleeding.

Statistical analysis will compare event-free survival of patients in 4 groups. Patients will be censored at the time of the occurrence of a kidney transplant, a dialysis method of change, a dialysis withdrawal, a move outside Lorraine, or date point if they are still alive . To minimize bias maximum indication, patients of different groups will be matched on propensity score (probability for a given patient to be treated by antiplatelet and / or anticoagulant).

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 and over,
* In end-stage renal disease,
* Initiating a first hemodialysis replacement therapy in Lorraine between 01/01/2009 and 31/12/2010.

Exclusion Criteria:

* Evolutionary Neoplasia at start of dialysis,
* Death within 45 days of the start of dialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for end-stage renal disease by chronic hemodialysis, in one of the 12 dialysis centers for adult Lorraine region (heavy or dialysis centers medicalized units).
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Survival without major clinical event | up to 54 months
  In Chronic Hemodialysis Patients

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie THILLY, Principal Investigator — n.thilly@chru-nancy.fr

IPD SHARING:
Plan to Share IPD: No